CLINICAL TRIAL: NCT06378073
Title: Effects of Chest Physiotherapy Exercise in Prevention of Pre-Operative and Post-Operative Complications Followed By Cardiac Surgery
Brief Title: Effects of Chest Physiotherapy Exercise in Prevention of Pre and Post Operative Complications By Cardiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/557
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Surgery-Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Spirometer (Experimental)
  Interventions: Diagnostic Test: Incentive Spirometer
- Numeric Pain Rating Scale (Other)
  Interventions: Diagnostic Test: Numeric Pain Rating Scale

INTERVENTIONS:
Diagnostic Test: Incentive Spirometer — Specificity and sensitivity: Incentive spirometry is a specific type of spirometry that aims to encourage people to breathe deeply intentionally but does not provide a measurement or inform management of chronic lung diseases. Less than 5 repetitions per day (sensitivity 93%, specificity 77%) and less than 2 balls per repetition (sensitivity 93%, specificity 77%) were predictive of postoperative pulmonary complications. (1) Validity and reliability: Incentive spirometry can be used as a simple mean to follow lung function, especially VC, in the postoperative period in spontaneously breathing patients. Incentive spirometry is noninvasive and can be performed repeatedly at the bedside in the intensive care setting. (2)
  Interpretation:
  There are only three numeric values that are required to interpret spirometry:
  * Forced Vital Capacity (FVC)
  * Forced Expiratory Volume (FEV1)
  * FEV1/FVC ratio.
  Arms: Incentive Spirometer
Diagnostic Test: Numeric Pain Rating Scale — Sensitivity: The area under the receiver operator characteristic curve for the NRS as a test for pain that interferes with functioning was 0.76, indicating fair accuracy. A pain screening NRS score of 1 was 69% sensitive for pain that interferes with functioning. (4) he diagnostic value of different NRS cut-off values for administering analgesics is determined by an ROC curve. Sensitivity of NRS > 3 for 'unbearable' pain in older patients was 72% with a specificity of 97·2%. With a cut-off point NRS > 4, sensitivity increased to 83%, while specificity was 96·7%. (5) Validity and reliability: The numerical rating scale is a reliable and valid tool for pain assessment in patients with musculoskeletal impairments. (3)
  Measurement (circle): Categorical /Numerical /Both:
  Numerical:
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
  Arms: Numeric Pain Rating Scale

SUMMARY:
"A randomized control trial will be conducted among 189 patients who have undergone cardiac surgery in past. The participants for this research will be patients of Pakistan Institute of Cardiology, University of Lahore Teaching Hospital, Azra Naheed Medical College and Bahria International Hospital. The chest physiotherapy technique will be applied on 2 controlled groups.

In 94 patients the effects of chest physiotherapy will be checked post - operatively and the effects will be checked on other half pre - operatively. The data will be gathered on practical performance and treatment based along with questionnaire. The data collected will then be analyzed using SPSS"

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing in Cardiac Surgery like, CABG, univalve, bivalve and trivalve.

Exclusion Criteria:

* Valve and CABG surgery combined with other cardiac surgery like percutaneous valve replacement.
* Cognitive disorder of the heart.

Ages: 48 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Incentive Spirometer | 6 Month
  A pain screening NRS score of 1 was 69% sensitive for pain that interferes with functioning. (4) Specificity: The diagnostic value of different NRS cut-off values for administering analgesics is determined by an ROC curve. Sensitivity of NRS > 3 for 'unbearable' pain in older patients was 72% with a specificity of 97·2%. With a cut-off point NRS > 4, sensitivity increased to 83%, while specificity was 96·7%. (5) Validity and reliability: The numerical rating scale is a reliable and valid tool for pain assessment in patients with musculoskeletal impairments.
Incentive Spirometer | 6 Months
  Specificity and sensitivity: Incentive spirometry is a specific type of spirometry that aims to encourage people to breathe deeply intentionally but does not provide a measurement or inform management of chronic lung diseases. Less than 5 repetitions per day (sensitivity 93%, specificity 77%) and less than 2 balls per repetition (sensitivity 93%, specificity 77%) were predictive of postoperative pulmonary complications.

CONTACTS AND LOCATIONS:
Locations (5):
- Pakistan (5):
  - Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - Bahria Hospital, Lahore, Punjab Province
  - Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - The University of Lahore Teaching Hospital, Lahore, Punjab Province
  - Punjab Institute of Cardiology Hospital, Lahore

IPD SHARING:
Plan to Share IPD: No